CLINICAL TRIAL: NCT01824719
Title: a Study of Clinical Safety Monitoring and the Mechanism of Anaphylactic Reaction Used Reduning(a Chinese Medicine Injection)in Hospitals in China
Brief Title: A Registry Study on Reduning（a Chinese Medicine Injection）Used in Hospitals in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yanming Xie, Director, China Academy of Chinese Medical Sciences
Other Study IDs: 200907001-5-6-1
Record Dates: First submitted 2013-03-30; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Upper Respiratory Tract Infection;; Acute Tracheobronchitis
MeSH Terms: conditions — Respiratory Tract Infections; Bronchitis

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Allergic group: All patients who used Reduning Injection have anaphylaxis.
- Control group: All patients who used Reduning Injection don't have anaphylaxis.One allergic group patient should matched four control group patients.

SUMMARY:
This study was advocated by Institute of Basic Research in Clinical Medicine, China Academy of Chinese Medical Sciences in January 2013.

The purpose of this study is to make a event monitoring to see whether Reduning injection is safe and the characteristic and mechanism of anaphylactic reaction used Reduning injection in hospitals in China.

DETAILED DESCRIPTION:
It is very common that Chinese Medicine Injection used in hospitals in mainland China. However safety problems rose in recent years. There could be many uncertain factors influence Chinese Medicine Injection in clinical practice.

In order to ensure the safety of public drug use and lower drug-induced risks, a registry study for Reduning injection safety surveillance with 3000 patients will be conducted from Jan.2013 to Mar.2013.At the same time,Patients who have anaphylactic reaction are selected as the allergic group and not have anaphylactic reaction are selected as the control group.The proportion of allergic group and control group is 1:4.All the patients who are selected should draw blood.

Eligibility criteria Patients who will use Reduning injection in selected hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients using Reduning injection from January to March 2013

Exclusion Criteria:

-

Ages: 1 Month to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An anticipated sample size was caculated in this study, about 3000 Patients using Reduning injection from January to March 2013 in hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with anaphylactic reaction;the blood routine examination of participants with anaphylactic reaction | to assess Reduning's 'anaphylactic reaction' .during patients' hospital stay, administration information of Reduning will be registered every day. The registry procedure will last 3 month only for patients using Reduning

CONTACTS AND LOCATIONS:
Overall Officials: Xie Y Ming, Principal Investigator — China Academy of Chinese Medical Sciences
Locations (1):
- Institute of Basic Research in Clinical Medicine, Beijing, Beijing Municipality, China